CLINICAL TRIAL: NCT06519071
Title: Determining Dietary Tryptophan Requirements In Healthy Pregnant Women Using The Indicator Amino Acid Oxidation Method
Brief Title: Tryptophan Requirements During Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Rajavel Elango, PhD, Principal Investigator, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: H23-01187
Record Dates: First submitted 2023-08-02; First posted 2024-07-25 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Pregnancy
Keywords: Amino Acids; Tryptophan; Pregnancy; Indicator Amino Acid Oxidation; Stable Isotopes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tryptophan Intake (Experimental): Randomly assign the participant to receive a test tryptophan oral intake (ranging between 1 to 14 mg.kg.d) as an 8-hourly isocaloric and isonitrogenous meal that consist of a liquid formula shake and protein-free cookies.
  Interventions: Other: Tryptophan Intake

INTERVENTIONS:
Other: Tryptophan Intake — Each hourly meal will provide one-twelfth of the participants' daily energy requirements as estimated by 1.7 Resting Energy Expenditure and adequate protein (at 1.5 g.kg.d), to maintain a metabolic steady state. The liquid shake contains protein-free powder orange-flavored drink crystals, corn oil, and water.

SUMMARY:
Pregnancy is an important period of life where there is an increased need for nutrients including protein and amino acids from food. The current protein and amino acids dietary recommendations were all established using older methods done in adult men. Then protein and amino acids requirements for all stages of pregnancy were calculated without accounting for changing demands in each trimester. Therefore, another more precise method is needed to better understand how much amino acids (in this study tryptophan) women need during pregnancy.

In the current study, the investigators are going to apply the Indicator Amino Acid Oxidation (IAAO) method to measure the dietary tryptophan needs in a healthy pregnancy. This method is a noninvasive, quick, and reliable technique that uses a stable isotope-labeled amino acid. The stable isotope tracer is a labeled amino acid, which is colorless, odorless, tasteless, and completely safe; they are present in the air, water and food. Amino acids are mostly made of Carbon-12 (12C), whereas the isotope tracer contains Carbon-13 (13C). The tracer can be detected in breath and urine samples with special equipment because it looks different than the rest of the amino acids in the body. In Elango lab, the investigators have done similar studies, using the same technique in children, nonpregnant women and pregnant women. This will allow us to measure tryptophan needs in pregnancy.

DETAILED DESCRIPTION:
Pre-Study:

All participants will arrive following a 10-12 hrs overnight fasting, to allow the anthropometric measurements, biochemical, and dietary assessments. Fasting blood glucose by finger prick will be used to screen for gestational diabetes. The presence of protein, glucose, ketones, leukocytes, and blood in urine will be assessed using urinalysis strips as potential indicators of gestational diabetes and preeclampsia. For the anthropometric assessment, weight and height will be measured and body composition will be determined using skinfold thickness measurements and Bioelectrical Impedance Analysis (BIA). A brief medical history will be obtained to screen for medication use, substance use, previous pregnancies, and overall health. For the dietary assessment, energy requirements will be determined using Resting Energy Expenditure (REE) by continuous, open-circuit indirect calorimetry. In addition to two-days detailed dietary records to estimate participants' calorie, protein, and tryptophan intake.

Study Day:

Participants are expected to arrive following a 10-12 hrs overnight fasting, as mentioned above, anthropometric measurements, fasting blood glucose testing and urine strip analysis will be repeated at the beginning of each study day. On the study day, the investigator will randomly assign the participant a test tryptophan intake (ranging between 1 to 14 mg.kg.d) and will receive an 8-hourly isocaloric and isonitrogenous meal. Based on Resting Energy Expenditure determined during the pre-study day, each meal will provide daily adequate energy and adequate protein (at 1.5 g.kg.d) to ensure that the Indicator Amino Acid Oxidation (IAAO) response is due to the different test tryptophan intakes and not from the limited energy and/or protein. During the study days, participants will be allowed to have the prepared study diets and water only.

Sample Collection:

Three baseline breath samples will be collected at 45, 30, and 15 min before isotope infusion. Thereafter isotope administration (meal 5 - 8), breath samples will be collected at 150, 180, 195, 210, 225, and 240 min during the metabolic steady state. Urine samples will be collected at 45 min before isotope infusion (meal 5) and two samples at 180, and 240 min after the tracer infusion. One blood sample will be collected to measure tryptophan and four related metabolites within the kynurenine and serotonin pathway (plasma kynurenine, xanthurenic acid, quinolinic acid, and serotonin), and B vitamins (plasma B6, B12, and B9) then compared between early and later stages of gestation in response to different tryptophan intakes.

ELIGIBILITY:
Inclusion Criteria:

* Cis-gendered pregnant woman.
* 20-40 years of age.
* Pregnant with a single child.
* Between 11-20 weeks of gestation or 31-40 weeks of gestation.
* Free of chronic diseases/acute diseases and have a full range of physical mobility.

Exclusion Criteria:

* Women who are not pregnant.
* Women who are pregnant with more than one child (this changes amino acid demands) or were pregnant in the 6 months before the current pregnancy.
* Women with a history of spontaneous abortion (within the last 6 months) or preterm birth.
* Women not in good health or have a metabolic, cardiovascular, neurological, genetic, or immune disorder, including gestational diabetes, preeclampsia, pregnancy-related anemia, or pregnancy-related jaundice.
* Claustrophobic women (a clear hood will be placed, which can easily be removed, over the participants head for approximately 20 min to measure energy expenditure).
* Women who are substance dependent (i.e., alcohol, tobacco, illicit drugs).
* Women who have severe nausea/vomiting throughout their pregnancy.
* Women under the age of 20 years and over the age of 40 years.
* Women who have lost weight (approximately 1.5kg or more) during their current pregnancy.
* Women with a pre-pregnancy Body Mass Index (BMI) under 19 or over 28 〖kg/m〗^2.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Cis-women.
Enrollment: 29 (Actual)
Dates: Start 2023-07-20 (Actual); Primary Completion 2025-03-20 (Actual); Study Completion 2025-07-18 (Actual)

PRIMARY OUTCOMES:
Carbon 13 Oxidation | 8 hours
  Urine and breath will be collected to measure the rate of oxidation of L-[1-13C]phenylalanine oxidation.

CONTACTS AND LOCATIONS:
Overall Officials: Rajavel Elango, PhD, Principal Investigator — University of British Columbia
Locations (1):
- BC Children's Hospital Research Institute, University of British Columbia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No